CLINICAL TRIAL: NCT05572151
Title: Determining the Optimal Examined Lymph Node for Accurate Staging and Long-term Survival in Rectal Cancer: a Population Study of the US Database and a Chinese Multi-institutional Registry
Brief Title: Determining the Optimal Examined Lymph Node for Accurate Staging and Long-term Survival in Rectal Cancer
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Shuai Jiao, Principal Investigator, The Second Affiliated Hospital of Harbin Medical University
Other Study IDs: 82100598
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lymph node number — Lymph nodes were harvested during surgical resection of rectal cancer

SUMMARY:
A multi-institutional registry of collected data on patients with rectal cancer who underwent surgical resection between January 2009 and December 2018 at the departments of colorectal surgery of five medical institutions in China

DETAILED DESCRIPTION:
A multi-institutional registry of collected data on patients with rectal cancer who underwent surgical resection between January 2009 and December 2018 at the departments of colorectal surgery of five medical institutions in China (National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Changhai Hospital, Naval Medical University; The Second Affiliated Hospital of Harbin Medical University; The Affiliated Tumor Hospital of Harbin Medical University; The Affiliated Tumor Hospital of Guangxi Medical University)

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer patients in stage I-III who underwent surgical resection for first primary rectal cancer with at least one lymph node were eligible

Exclusion Criteria:

* Patients with missing values on lymph node count and clinical features were excluded

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Information about patients (age, sex and year of diagnosis), tumor (TNM stages, histology, size and differentiation), treatments (resection type, chemotherapy), and outcome variables (follow-up time and survival status) were obtained in SEER database and China registry
Sampling Method: Probability Sample
Enrollment: 7694 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
lymph node number | during the surgery
  lymph nodes were harvested during surgical resection of rectal cancer

REFERENCES:
- [Background] Del Paggio JC, Peng Y, Wei X, Nanji S, MacDonald PH, Krishnan Nair C, Booth CM. Population-based study to re-evaluate optimal lymph node yield in colonic cancer. Br J Surg. 2017 Jul;104(8):1087-1096. doi: 10.1002/bjs.10540. Epub 2017 May 24. PMID 28542954
- [Derived] Guan X, Jiao S, Wen R, Yu G, Liu J, Miao D, Wei R, Zhang W, Hao L, Zhou L, Lou Z, Liu S, Zhao E, Wang G, Zhang W, Wang X. Optimal examined lymph node number for accurate staging and long-term survival in rectal cancer: a population-based study. Int J Surg. 2023 Aug 1;109(8):2241-2248. doi: 10.1097/JS9.0000000000000320. PMID 37428195